CLINICAL TRIAL: NCT04766606
Title: Management of Anticoagulant Therapy in Non-cardiac Surgical Patients in Relation to Their Postoperative Clinical Outcome.
Brief Title: Management of Anticoagulant Therapy in Non-cardiac Surgery.
Status: Completed | Type: Observational
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, BOLOSI MARIA, Consultant Anaesthesiologist, University of Ioannina
Other Study IDs: 609a/25-11-2019
Record Dates: First submitted 2021-02-14; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Antithrombotic Agents Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The perioperative treatment of patients receiving long-term anticoagulant therapy is challenging. This is attributed to the continuation of anticoagulants perioperatively, which is associated with an increased bleeding risk while their discontinuation increases the risk of thromboembolic or ischemic events.

Type of surgery and patient's comorbidities (i.e. haematological diseases, renal or hepatic insufficiency, and concomitant use of other anticoagulants) are significant factors associated with perioperative bleeding. Bleeding risk is stratifies according to the 2011 Canadian Cardiovascular Society Guidelines for the Management of Patients with Antiplatelet Disorder. Surgical thrombotic risk assessment is based on 2014 ESC / ESA Guidelines on non-cardiac surgery.

The purpose of this study is to investigate and record the management of anticoagulant therapy and long term outcome. The primary target is to record the anticoagulant management in non-cardiac elective surgery during one year in our Hospital. The study involves the investigation of the degree of compliance according to published guidelines. Immediate postoperative complications and major events are secondary goals. Data are assessed at 30, 90 days and one year follow up after surgery.

Understanding the need to discontinue or not antithrombotic agents and adapting treatment strategies according to type of surgery is the key to balance their safety and efficacy. Cardiologists, surgeons, and anaesthesiologists should be aware of the potential catastrophic risks of early discontinuation or continuation of antithrombotic therapy.

DETAILED DESCRIPTION:
It is estimated that more than 150,000 patients receive anticoagulant treatment in Greece. More than 10% of those will need to undergo surgery annually. Major side effects of all anticoagulants are bleeding or major thromboembolic events perioperatively.

The perioperative treatment of patients receiving long-term anticoagulant therapy is challenging. This is attributed to the continuation of anticoagulants perioperatively, which is associated with an increased bleeding risk while their discontinuation increases the risk of thromboembolic or ischemic events.

Type of surgery and patient's comorbidities (i.e. haematological diseases, renal or hepatic insufficiency, and concomitant use of other anticoagulants) are significant factors associated with perioperative bleeding. According to the 2011 Canadian Cardiovascular Society Guidelines for the Management of Patients with Antiplatelet Disorder, bleeding risk is stratified as following:

* Very high risk: neurosurgery (intracranial or spinal surgery), cardiac surgery (coronary artery bypass grafting or valve replacement).
* Medium risk: intrathoracic, intra-abdominal procedures, orthopaedic, vascular and other selective procedures (prostate or cervical biopsy).
* High Risk: major vascular surgeries (abdominal aortic aneurysm, aortic bypass), major orthopaedic surgery on the lower extremity (total hip / knee), pneumonectomy, enterectomy, placement of permanent pacemaker or internal defibrillator and other selected procedures (kidney biopsy, pericardium puncture, resection of colon polyps).
* Low risk: laparoscopic procedures (cholecystectomy, inguinal hernia repair), dental, dermatological, ophthalmic procedures, coronary angiography, gastroscopy /colonoscopy and other selected procedures (bone marrow or lymph node biopsy, thoracotomy, joint puncture).
* Very low risk: low risk dental procedures (i.e. tooth extraction), skin biopsy or skin cancer excision, cataract surgery.

Surgical thrombotic risk assessment is based on 2014 ESC / ESA Guidelines on non-cardiac surgery. Low risk (<1%) surgeries include superficial surgery, breast procedures etc., medium risk (1-5%) splenectomy, cholecystectomy, etc., and high risk (>5%) are major aortic and other major blood vessel operations, open limb revascularization or amputation or embolectomy, gastric surgery, hepatectomy, etc.

The purpose of this study is to investigate and record the management of anticoagulant therapy and long term outcome. The primary target is to record the anticoagulant management in non-cardiac elective surgery during one year in our Hospital. The study involves the investigation of the degree of compliance according to published guidelines. Immediate postoperative complications and major events are secondary goals. Data are assessed at 30, 90 days and one year follow up after surgery.

Data recording involves patient demographics, somatometric data, medical history, comorbidities and home medication. Specifically, details concerning antiplatelet or anticoagulant medication, such as diagnosis, duration of treatment, time to treatment discontinuation prior surgery, bridging, intraoperative administration of anticoagulants if needed, time of re-administration postoperatively and what medical specialties were involved in the perioperative management of antithrombotic agents are also included. Hospital length of stay is also recorded. Complications recorded during the one year study period include the following: acute myocardial infarction, pulmonary embolism, vascular haemorrhage, sudden death, arrhythmias, aneurysm rupture, bleeding and management, and other major events. Moreover, after patient discharge, all cause re-hospitalization and any alteration to antithrombotic treatment is also recorded.

Perioperative management of patients receiving antithrombotics is multifactorial and high quality evidence is lacking. The achievement of the delicate balance between efficacy and safety, between thrombotic and hemorrhagic risk, remains a challenge for the physicians who are called upon to treat patients under antithrombotic agents who are candidates for surgery. Understanding the need to discontinue or not antithrombotic agents and adapting treatment strategies according to type of surgery is the key to balance their safety and efficacy. Cardiologists, surgeons, and anaesthesiologists should be aware of the potential catastrophic risks of early discontinuation or continuation of antithrombotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* non-cardiac surgery
* general, urological, orthopaedic, gynecological, ophthalmological, ENT, plastic surgery and neurosurgery

Exclusion Criteria:

* age under 18 years old
* emergency surgery
* mental disorders
* caesarean sections
* surgeries lasting less more than 20 minutes
* patients' refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients submmitted for elective non cardiac surgery in University Hospital of Ioannina during one year period.
Sampling Method: Non-Probability Sample
Enrollment: 614 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Perioeprative antithrombotic management in elective non-cardiac elective surgery. | One weak prior to surgery until one year follow up.
  Recording of cause of antithrombotic therapy ( ICD-10).
Perioeprative antithrombotic management in elective non-cardiac elective surgery. | One weak prior to surgery until one year follow up.
  Recording of type of preoperative antithrombotic agent (description of treatment).
Perioeprative antithrombotic management in elective non-cardiac elective surgery. | Perioperatively (one week before surgery until 30 days after surgery).
  Recording of need of bridging therapy (yes or no).
Perioeprative antithrombotic management in elective non-cardiac elective surgery. | Postoperatively (until 30 days after surgery).
  Recording time of re-administration of antithrombotic therapy postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: Undecided